CLINICAL TRIAL: NCT05120310
Title: Testing the Effects of the Calm App on Sleep, Mental Health, and Productivity Outcomes in Employees
Brief Title: Effects of Health and Wellness App on Employee Productivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00014072
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sleep Disturbance; Mental Health Wellness 1
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: There will be two groups: first is the intervention group and the other is a waitlist-control and will receive the intervention after the control portion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be asked to use the Calm app for at least 10 minutes per day for eight weeks. They will also be asked to schedule one live 20-minute coaching session with a Calm Coach within the first week of the eight-week intervention to help identify areas for health behavior improvements (i.e., Calm Concierge).
  - Calm Coaching for sleep Subsample (N=100): A random subsample of eligible participants, based on their ISI scores, will be invited to use the Calm Coaching for Sleep Program (using Healthie platform).
  Interventions: Behavioral: The Calm App
- Waitlist Control (Other): Participants will be instructed to not participate in any mindfulness meditation activities for eight weeks. The research team will send the participant study instructions. At the end of eight weeks participants will be given access to the Calm app and will be able to schedule one live 20-minute coaching session with a Calm Coach.
  - Calm Coaching for sleep Subsample (N=100): A random subsample of eligible participants, based on their ISI scores, will be invited to use the Calm Coaching for sleep Program. The Calm Coaching for sleep program is administered by Calm for six weeks.
  Interventions: Behavioral: The Calm App

INTERVENTIONS:
Behavioral: The Calm App — Participants will be asked to use the Calm app for at least 10 minutes per day for eight weeks. They will also be asked to schedule one live 20-minute coaching session with a Calm Coach within the first week of the eight-week intervention to help identify areas for health behavior improvements (i.e., Calm Concierge). Participants will be asked to download the Calm app to their mobile phone. The Calm Coaching for sleep program is administered by Calm for six weeks. Participants are asked to complete weekly modules and interact with a coach to help them improve their sleep. Participants also complete a sleep diary throughout the program.

SUMMARY:
The purpose of this study is to test the effects of using the Calm app + coaching concierge (one 20-min session) and/or Calm Coaching for sleep program on sleep, mental health, and work productivity outcomes in employees.

Employees (N=5,000) will be randomized into one of two groups for 8-weeks.

DETAILED DESCRIPTION:
Workplace stress is highly prevalent and is linked to poor health outcomes including depression and anxiety. Depression impacts a person's physical ability to complete job tasks about 20% of the time while reducing cognitive performance 35% of the time. Mental health issues are not often properly identified and less than half of people receive treatment.

The Calm app is a mindfulness meditation mobile app and has been evidenced to reduce stress, improve sleep, and reduce anxiety/depressive symptoms in a range of populations (e.g., college students, cancer patients, sleep-disturbed adults). The Calm app provides daily, 10-minute, guided meditations grounded in mindfulness-based stress reduction (MBSR) and Vipassana meditation. Uniquely, the Calm app also offers "Sleep Stories", narrated fictional tales that use mindfulness- inspired techniques to help users sleep. However, the effects of the Calm app in employees among worksites has not yet been explored.

The purpose of this study is to test the effects of using the Calm app + coaching concierge (one 20-min session) and/or Calm Coaching for sleep program on sleep, mental health, and work productivity outcomes in employees.

Employees (N=5,000) will be randomized into one of two groups for 8-weeks.

The research team will randomize the employee sites into one of two groups

1. Intervention group (N=2,500): Calm app + concierge (one live 20-minute coaching session)

   a. Calm Coaching for sleep Subsample (N=100): Participants with elevated sleep disturbance (determined as a score of >10 with the ISI) AND interest in Calm Coaching for sleep will be assigned to the Calm Coaching for sleep Program in addition to having the Calm app + concierge
2. Waitlist control group (N=2,500): Following 8-weeks from the study start date, employee receives access to the Calm app a. Calm Coaching for sleep Subsample (N=100): Participants with elevated sleep disturbance (determined as a score of >10 with the ISI) AND interest in Calm Coaching for sleep will be assigned to the Calm Coaching for sleep Program in addition to having the Calm app + concierge

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Employee of company
* Only English speakers
* Willing to download the Calm app to their smartphone

Exclusion Criteria:

• Greater than 60 minutes/month of meditation for the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | Change from baseline daytime sleepiness at 8-weeks; 8-items; Scores range from 0-24 with higher scores indicating higher levels of daytime sleepiness.
  Daytime sleepiness
Insomnia Severity Index | Change from baseline symptoms of insomnia at 8-weeks; 7-items; Scores range from 0-28 with higher scores indicating greater symptoms of insomnia.
  Symptoms of insomnia

SECONDARY OUTCOMES:
Pittsburgh Sleep Diaries | Daily for 6 weeks
  Sleep diaries assessing sleep/wake time and sleep quality
Productivity | Change from baseline to post-intervention (week 8)
  Productivity will be measured using the Work Productivity and Activity Impairment Questionnaire. Scores on the WPAI:GH are provided as a percentage with higher numbers indicating greater impairment and less productivity.
Resilience | Change from baseline to post-intervention (week 8)
  Resilience will be measured using the Brief Resilience Scale, with scores ranging from 1-5, and a higher score indicates a better outcome.
Depression, Anxiety, and Stress Scale | Change from baseline to post-intervention (week 8)
  Depression, Anxiety, and Stress Scale will be measured using the Depression, Anxiety, and Stress Scale (DASS-21) with lower scores in the three categories indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espel-Huynh H, Baldwin M, Puzia M, Huberty J. The Indirect Effects of a Mindfulness Mobile App on Productivity Through Changes in Sleep Among Retail Employees: Secondary Analysis. JMIR Mhealth Uhealth. 2022 Sep 28;10(9):e40500. doi: 10.2196/40500. PMID 36169994
- [Derived] Huberty JL, Espel-Huynh HM, Neher TL, Puzia ME. Testing the Pragmatic Effectiveness of a Consumer-Based Mindfulness Mobile App in the Workplace: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Sep 28;10(9):e38903. doi: 10.2196/38903. PMID 36169991